CLINICAL TRIAL: NCT04456972
Title: Pilot Study on the Contribution of Molecular Analysis of Endometrial Cancers: Reliability, and Interest of Circulating Tumor DNA
Brief Title: Reliability and Interest of Circulating Tumor DNA in Endometrial Cancers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ENDOCIRC
Record Dates: First submitted 2020-06-15; First posted 2020-07-07 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Circulating Tumor DNA; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm only (Experimental)
  Interventions: Diagnostic Test: One arm only

INTERVENTIONS:
Diagnostic Test: One arm only — Samples of plasma to analyze ctDNA

SUMMARY:
The recent histo-prognostic molecular discoveries of the TCGA (The Cancer Genome Atlas) have shed new light on the classification of endometrial carcinomas.

After carrying out different types of high-throughput molecular analyzes on 373 endometrial carcinomas of different histological types, 4 major tumor subtypes could be identified, each with a different survival profile (the "ultra-mutated" group with POLE mutations, the "hypermuted" group with microsatellite instability (MSI), the "low number of copies" group, and the "high number of copies" group).

This histomolecular classification is not yet directly transposable to clinical practice and tumor genetic characteristics have not had any direct therapeutic impact to date.

The main objective of the study is to determine the concordance rate between molecular analysis of tumor tissue and that of cDNA in patients with endometrial cancer during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven endometrial adenocarcinoma type I or type II.
* With recent abdomino-pelvic imaging, less than 3 months old.
* Tumor tissue sufficiently exploitable for research (> 20% of tumor cells)
* Informed consent signed by the patient after clear and fair information about the study.
* Free patient, without tutorship, curatorship or subordination.
* Patient benefiting from a Social Security scheme or benefiting from it through a third person.
* Patient not opposed to participating in the study.

Exclusion Criteria:

* Histologies other than adenocarcinoma (sarcoma, leiomyosarcoma)
* Linguistic or mental refusal or incapacity to understand and / or sign the informed consent
* Patients benefiting from enhanced protection, namely: minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection.
* Pregnant and / or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to determine the concordance rate between molecular analysis of tumor tissue and that of cDNA in patients with endometrial cancer during treatment. | 15 days
  Concordance between molecular analysis of tumor tissue and that of cDNA, in patients with endometrial cancer during treatment

SECONDARY OUTCOMES:
Analysis of the association of molecular anomalies on cDNA with clinical histological data. | 15 days
  Association of molecular analyzes of tumor tissue DNA with clinical and histological data available at inclusion.
Analysis of the association of molecular anomalies on cDNA and the amount of total circulating DNA to the radiological response in a metastatic situation. | 3 months
  Association of the detection of molecular anomalies from cDNA, and the amount of total circulating DNA, with the radiological response in the metastatic population.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Mrs EVRARD, PHD, Principal Investigator — CHU Poitiers
Locations (1):
- CHU Poitiers, PRC, Poitiers, France

IPD SHARING:
Plan to Share IPD: No
Analyzes will be only realised on biology molecular plateform at CHU Poitiers on a first time.
  If we failed to obtain results we perhaps send plasma in other laboratory